CLINICAL TRIAL: NCT06113120
Title: Specific Role of Nurse in a Mobile Palliative Care Team (EMSP): Real Autonomy or Utopia
Acronym: AutonInfSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8901
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-10

CONDITIONS: Palliative Care
Keywords: Improving patients care; Nurse; Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A bibliographic search carried out by the investigators demonstrated that there are few studies or data relating to the role and place of a State Registered Nurse (IDE) in a Mobile Palliative Care Team (EMSP) concerning the collection and the analysis of the needs expressed when formulating an evaluation request by the EMSP. The IDE collects, questions, analyzes needs and initiates an evaluation with the patient or, failing that, advises and/or redirects. This first necessary step before the overall evaluation led the investigators to question the autonomy of the IDE in an EMSP and to research what are the representations of an IDE in this role of collecting and analyzing needs. when making such a request?

The aim of this research is to explore the professional practices of nurses within other PMSCs in order to analyze them and move towards improving patient care.

ELIGIBILITY:
Inclusion criteria:

* State-certified nurse working in EMSP with intra- and extra-hospital activity in a CHRU or CHU.
* Subject having given their consent for the reuse of their data for the purposes of this research

Exclusion criteria:

* Subject having expressed opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: State-certified nurse working in EMSP with intra- and extra-hospital activity in a CHRU or CHU.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03-09 (Estimated)

PRIMARY OUTCOMES:
Review of professional practices in Palliative Care | Study covers the period from February 9, 2023 to March 9, 2024
  The study consisted of an inventory of professional practices of nurses within mobile palliative care teams

CONTACTS AND LOCATIONS:
Locations (1):
- Service de soins Palliatifs - CHU de Strasbourg - France, Strasbourg, France